CLINICAL TRIAL: NCT05538910
Title: Defining Neurobiological Links Between Substance Use and Mental Illness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 10000922; 000922-DA
Record Dates: First submitted 2022-09-08; First posted 2022-09-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01-16

CONDITIONS: Major Depressive Disorder; Substance Use Disorder; Normal Physiology
Keywords: fMRI; Reward Function; Affective Processing; Interoceptive Awareness
MeSH Terms: conditions — Depressive Disorder, Major; Substance-Related Disorders | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Placebo (Placebo Comparator): Placebo patch + Placebo Pill
  Interventions: Other: Placebo Nicotine Patch
- Arm 2: Nicotine Patch (Experimental): Nicotine Patch + Placebo Pill
  Interventions: Drug: Nicotine Patch

INTERVENTIONS:
Other: Placebo Nicotine Patch — Comparator
  Arms: Arm 1: Placebo
Drug: Nicotine Patch — Study drug: 7.5 mg Nicotine Patch which will be administered in a double blind, randomized manner
  Arms: Arm 2: Nicotine Patch

SUMMARY:
Background:

Nicotine dependence leads to about 480,000 deaths every year in the United States. People with major depressive disorder (MDD) are twice as likely to use nicotine compared to the general population. They have greater withdrawal symptoms and are more likely to relapse after quitting compared with smokers without MDD. More research is needed on how nicotine affects brain function in those with MDD.

Objective:

To understand how nicotine affects symptoms of depression and related brain function.

Eligibility:

People aged 18 to 60 years, at the time of consent, with and without MDD who do not smoke cigarettes or use other nicotine products.

Design:

Participants will have 2 or 3 study visits over 1 year.

Participants will have 2 MRI scans no less than 4 days apart. Each scan visit will last 5 to 7 hours. At each scan, they will have urine and breath tests to screen for recent use of alcohol, nicotine, and illegal drugs.

Before each scan, they will take 1 of 2 medications: nicotine or placebo. Participants will receive each medication once. They will not know which medication they are receiving at each scan.

For each MRI scan, they will lie on a table that slides into a cylinder. Sometimes they will be asked to lie still. Sometimes they will complete tasks on a computer. Tasks may include identifying colors or playing games to win money. Each scan will take about 2 hours.

Participants will answer questions about their thoughts, feelings, and behaviors before and after each scan.

They will have a blood test after each scan.

DETAILED DESCRIPTION:
Study Description:

Tobacco smoking leads to 480,000 deaths and a loss of $300 billion a year in the U.S. Individuals with major depressive disorder (MDD) are more vulnerable for experiencing these burdens as they are twice as likely to use nicotine versus the general population. The current work will explain the neurobiological basis of this enhanced risk and will define potential targets for lessening the impact of nicotine on those with MDD. This research plan will take the innovative approach of evaluating nicotine s effects in non-smokers with and without MDD. In contrast to focusing on nicotine dependent individuals, which introduces confounds due to chronic use, this design will directly show the domains in which the neurobiological impact of nicotine is greater in those with MDD, providing a mechanistic framework for enhanced risk.

To further characterize the links between nicotine use and mental illness, a second arm of the protocol will evaluate the impact of mental health comorbidities on the neurobiological impact of nicotine in individuals who use nicotine regularly. This secondary arm of the protocol will provide a more complete picture of why individuals with mental health comorbidities are at higher risk of nicotine dependence than the general population.

Objectives:

The primary objective of the first study arm is to determine the differential neurobiological impact of a nicotinic agonist on those with and without current major depressive disorder. Whether such effects are linked with specific symptoms of MDD will be assessed as will the potential modifying influence of biological sex. Those with a lifetime history of MDD will be assessed as well given evidence that reduced reward responsivity is a trait that persists even when one no longer meets current MDD criteria.

The primary objective of the second study arm is to determine the impact of nicotine-modulated changes in brain function, cognition, and affect between those who do and do not chronically use nicotine. Psychiatric symptoms will be evaluated along dimensions of internalizing (e.g., depression, anxiety), thought disorders (e.g. psychosis), and externalizing (e.g., impulsivity, ADHD) to characterize the full spectrum of mental health symptoms that may influence the neurobiological impact of nicotine.

Endpoints:

Brain function will be assessed in several ways: 1) Resting-state fMRI will determine pharmacologically mediated group-specific differences in functional brain organization and inherent dynamic functioning 2) Task-based fMRI will determine pharmacologically mediated group-specific differences in reward function, affective processing, and interceptive awareness. These same measures will further be assessed considering specific symptoms of MDD and biological sex.

In the arm of individuals using nicotine, brain function will be assessed using task and resting-state fMRI to determine the associations between mental health symptom dimensions and pharmacologically mediated associations with (1) functional brain organization and inherent dynamic functioning and (2) reward function, cue-reactivity, affective processing, and interoceptive awareness.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for this study, an individual must meet all the following criteria assessed under the currently approved NIDA IRP screening protocol for the evaluation of potential research subjects (here referred to as the NIDA screening protocol). This is a protocol led by the Office of the Clinical Director (OCD) at the National Institute on Drug Abuse Intramural Research Program (NIDA IRP) to assess potential research participants eligibility for entering clinical protocols at the NIDA/IRP. Additional details can be found in the NIDA screening protocol documents. As routinely done at the NIDA IRP, the screening procedures and data collected under the NIDA

screening protocol will capture information above and beyond what is necessary to determine eligibility for this protocol but allows the Investigators to assess the eligibility criteria for this protocol.

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

All Participants:

1. Able and willing to provide written informed consent.
2. Both sexes and all ethnic origins, age between 18 and 60 at the time of consent. Justification: Many neural processes change with age, and these changes could introduce unwanted variability in both behavioral and MRI signals.
3. Be generally healthy
4. Absence of pregnancy and breastfeeding. Justification: study procedures and drugs used in the current protocol may complicate pregnancy or be transferred to nursing children. Assessment tool(s): Urine and/or serum pregnancy tests, and clinical interview. Urine pregnancy tests will also be conducted at the beginning of each imaging visit.
5. Have a Breath Alcohol Value of 0 on all study visit days involving scanning. Participant may be rescheduled if this value is greater than 0.

MDD Subjects:

1. Meet DSM-5 diagnostic criteria for current MDD at screening Clinical judgement will be used to interpret criteria.
2. Have a baseline (Hamilton Depression) HAM-D score indicative of current depression as evaluated by clinical staff.
3. Current stable serotonin modulating drug (e.g. SSRI/SNRI/serotonin modulator) treatment is allowed (no changes in the last 2 months). Specific medications will be evaluated by the MAI.

Remitted MDD Subjects:

1. Meet DSM-5 diagnostic criteria for remitted MDD (full remission or partial remission or past depression) Clinical judgement will be used to interpret criteria.
2. HAM-D score indicating no clinically relevant depression as evaluated by clinical staff.
3. Current stable serotonin modulating drug (e.g. SSRI/SNRI/serotonin modulator) treatment is allowed (no changes in the last 2 months). Specific medications will be evaluated by the MAI.

Control Subjects (without MDD):

1. In addition to the absence of medical, neurological, and psychiatric illness listed above, control participants must not have current/lifetime MDD. Clinical judgement will be used to interpret criteria.
2. HAM-D score indicating no clinically-relevant depression as evaluated by clinical staff.

Daily Nicotine Users (Study Arm 2):

1. Uses nicotine daily for at least six months
2. Positive urine screen for cotinine

EXCLUSION CRITERIA (STUDY ARM 1):

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Subjects with suicidal ideation where outpatient treatment is determined unsafe.
2. Lifetime history or current diagnosis of any of the following psychiatric illnesses: organic mental disorder, schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorders not otherwise specified, bipolar disorder, patients with mood congruent or mood incongruent psychotic features. The MAI and/or PI/LI will reserve the right to exclude based psychiatric history not explicitly described in this criterion

   a. Within the control group, Current/lifetime MDD will be exclusionary for controls. Those currently using antidepressants to treat anxiety disorders typically co-morbid with MDD such as general anxiety disorder and panic disorder will be excluded. The MAI will reserve the right to exclude on the basis of psychiatric history not explicitly described in this criterion.
3. Are cognitively impaired or have a learning disability severe enough to have required intervention throughout most or all of K-12 education. The MAI will reserve the right to evaluate if a participant s history of educational placement is likely to represent a learning disability that could significantly impact the data gathered in this study based on the severity and type of learning disability. Justification: Cognitive impairment and learning disabilities may be associated with altered brain functioning in regions recruited during laboratory task performance.
4. Heavy caffeine users (consume greater than 500 mg on a regular or daily basis. This is approximately five 8 fl oz cups of coffee). Participants will be asked to not deviate from their typical caffeine use on all scanning days.
5. May not have regularly used any nicotine product in the past year; must never have been daily nicotine users for more than 1 month.
6. Must have an expired carbon monoxide level of less than or equal to 5 ppm and cotinine levels consistent with a non-smoker. Depending on the commercially available test used, a level equivalent to a non-smoker status will be used, ideally indicative of a urine cotinine level of around 10 ng/ml. However, given the known limitations of rapid tests to return specific quantifications of cotinine levels, if the present test is unable to quantify cotinine at this level, the lowest level of detection will be used as a cut off and MAI / PI discretion may be used to determine whether this cut off coupled with participant history and environmental factors indicates personal nicotine use versus secondhand smoke environment.
7. History of moderate or severe substance use disorder in the past 6 months (other than caffeine)
8. Current pharmacological treatment for opioid use disorder (i.e., use of methadone)
9. Current use of illegal drugs other than marijuana as measured by urine drug screen Marijuana will not be allowed in the 24 hours prior to scanning based on self-report. Study day can be rescheduled to accommodate.
10. Participants may not use anticholinergic drugs (i.e., scopolamine), dopamine enhancing drugs (i.e. methylphenidate), or other medications that may impact MRI measures (i.e. benzodiazepines) prior to any scanning visit within a timeframe that is likely to directly

    impact the study questions. MAI discretion regarding timeframe of allowed use will be based on half-life, pharmacology of the drug in question, and pattern of use by the participant. Scanning visit timing can be adjusted to accommodate.
11. May not use drugs that directly enhance dopamine (i.e., methylphenidate) in the week prior to any scanning visit. Scanning visit timing can be adjusted to accommodate.
12. Any past or present significant cardiovascular, cerebrovascular, or respiratory conditions, including arrhythmias, acute coronary syndrome, ischemic heart disease, or, uncontrolled hypertension
13. Body mass index (BMI) lower than 18.5 kg/m^2
14. Contraindications to MRI as determined by MRI Safety Screening form and mock scanner trial (when available).
15. Abnormal structural MRI, significant head trauma, current neurological illness including but not limited to frequent migraines, multiple sclerosis, movement disorder
16. Lifetime history of significant seizure disorder
17. Any other serious or unstable medical illness as defined by self-report, the evaluation of vital signs or other observation that in the view of the investigators would compromise the safety of an individual during participation

    All data collected will be evaluated by members of the study team to decide if there is an existing medical illness that would compromise participation in this research
18. Subjects that cannot speak English. Justification: To include non-English speakers, we would have to translate the consent and other study documents and hire and train bilingual staff, which would require resources that we do not have and could not justify, given the small sample size for each experiment. Additionally, the data integrity of some of the cognitive tasks and standardized questionnaires used in this study would be compromised as they have only been validated in English. Most importantly, ongoing communication regarding safety procedures is necessary when participants are undergoing MRI procedures. The inability to effectively communicate MRI safety procedures in a language other than English could compromise the safety of non-English speaking participants

Exclusion Criteria (Study Arm 2)

1. Subjects with active suicidal ideation where outpatient treatment is determined unsafe.
2. Current psychiatric symptoms in which the ability to adhere to study protocol is determined to be impaired by clinical staff/MAI (e.g., difficulty understanding or answering questions, difficulty remaining still in the fMRI scanner)
3. Are cognitively impaired or have a learning disability severe enough to have required intervention throughout most or all of K-12 education. The MAI will reserve the right to evaluate if a participant s history of educational placement is likely to represent a learning disability that could significantly impact the data gathered in this study based on the severity and type of learning disability.

   Justification: Cognitive impairment and learning disabilities may be associated with altered brain functioning in regions recruited

   during laboratory task performance.
4. Heavy caffeine users (consume greater than 500 mg on a regular or daily basis. This is approximately five 8 fl oz cups of coffee). Participants will be asked to not deviate from their typical caffeine use on all scanning days.
5. Active severe substance use disorder in the past 6 months (other than caffeine and nicotine)
6. Contraindications to MRI as determined by MRI Safety Screening form and mock scanner trial (when available).
7. Abnormal structural MRI, significant head trauma, current neurological illness likely to impact fMRI signal or ability to comply with study requirements (e.g., staying still in scanner)
8. Any serious or unstable medical illness as defined by self-report, the evaluation of vital signs or other observation that in the view of the investigators, would compromise the safety of an individual during participation. All data collected will be evaluated by members of the study team to decide if there is an existing medical illness that would compromise participation in this research
9. Subjects that cannot speak English. Justification: To include non-English speakers, we would have to translate the consent and other study documents and hire and train bilingual staff, which would require resources that we do not have and could not justify, given the small sample size for each experiment. Additionally, the data integrity of some of the cognitive tasks and standardized questionnaires used in this study would be compromised as they have only been validated in English. Most importantly, ongoing communication regarding safety procedures is necessary when participants are undergoing MRI procedures. The inability to effectively communicate MRI safety procedures in a language other than English could compromise the safety of non-English speaking participants

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 620 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
4.Nicotine effects and symptoms of MDD | At each scan visit
  Greater expression of MDD symptoms will related to a larger nicotine-induced impact within that domain.
3. Task and Resting State Brain | At each scan visit
  Relate static and temporal dynamic resting state brain function to nicotinic effects.
2.Task-fMRI | At each scan visit
  2. Evaluate nicotine agonism on: 1) different phases of reward processing, 2) brain/behavioral measures of attentional bias using the classic and emotional Stroop task, and 1.3. 3) interoceptive awareness. 4) confidence on value-based decisions, determine the influence of sex in the context of points 1-3.
1.Resting-fMRI | At each scan visit
  1.Determine the impact of nicotine agonism on the brain s inherent function and organization at rest.

SECONDARY OUTCOMES:
Determine the relationship between blood-based biomarkers, such as inflammatory makers/metabolomics and nicotinic effects | Ongoing
  Correlate levels of blood-based biomarkers with brain and behavioral measures and determine whether nicotine...

CONTACTS AND LOCATIONS:
Overall Officials: Amy C Janes, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share data as specified in the protocol and potentially through future data transfer agreement(s). Any shared data will be stripped of identifiers prior to release for sharing. De-identified data may be shared with properly administered databases and/or with collaborators with whom proper data sharing agreements are in place. Outside of the data sharing plan already specified in the protocol (in what would be outline in a future data sharing agreement), we have not yet finalized decisions on types of supporting information that will be shared, IPD Sharing Time Frame, IPD Sharing Access Criteria for other future data sharing agreements.